CLINICAL TRIAL: NCT06627712
Title: Stereotactic Body Radiotherapy (SBRT) Combined With PD-1 Inhibitor and Chemotherapy in Early-stage Treatment-naive Triple-negative Breast Cancer Patients: A Multicenter Phase III Clinical Study
Brief Title: SBRT Combined With PD-1 Inhibitor and Chemotherapy in Early-stage TNBC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20241776
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: Triple negative breast cancer; SBRT; Chemotherapy; PD-1 Inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT+PD-1 Inhibitor + Chemotherapy (Experimental): Radiotherapy: 24Gy/3f, once every other day; Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle; Carboplatin AUC=5, IV, administered on day 1 of each cycle.
  Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Interventions: Drug: SBRT+PD-1 Inhibitor + Chemotherapy
- PD-1 Inhibitor + Chemotherapy (Placebo Comparator): Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle; Carboplatin AUC=5, IV, administered on day 1 of each cycle.
  Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Interventions: Drug: PD-1 Inhibitor + Chemotherapy

INTERVENTIONS:
Drug: SBRT+PD-1 Inhibitor + Chemotherapy — Radiotherapy: 24Gy/3f, once every other day; Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle; Carboplatin AUC=5, IV, administered on day 1 of each cycle.
  Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Arms: SBRT+PD-1 Inhibitor + Chemotherapy
Drug: PD-1 Inhibitor + Chemotherapy — Chemotherapy: Cycles 1-4: Albumin-bound paclitaxel: 260 mg/m², IV, administered on day 1 of each cycle; Carboplatin AUC=5, IV, administered on day 1 of each cycle.
  Cycles 5-8: Epirubicin: 90-100 mg/m², IV, administered on day 1 of each cycle; Cyclophosphamide: 600 mg/m², IV, administered on day 1 of each cycle; Immunotherapy: PD-1 inhibitor, once every three weeks
  Arms: PD-1 Inhibitor + Chemotherapy

SUMMARY:
Triple-negative breast cancer (TNBC) presents significant challenges due to its limited treatment options and poor efficacy. While neoadjuvant chemotherapy has improved breast-conserving rates and extended survival for TNBC patients, this subtype still faces issues such as restricted treatment modalities, low pathological response rates, and unfavorable prognosis compared to other subtypes. Studies like Keynote522 and IMpassion031 have shown that combining chemotherapy with immunotherapy yields a pCR rate of 64.8% in early-stage high-risk TNBC patients, suggesting that such combinations can offer substantial benefits. However, the low immunogenicity of breast cancer and the lack of clear predictive molecular markers for effective immunotherapy result in suboptimal pCR and objective response rates for this group. Radiotherapy has systemic immune regulatory effects by promoting the release of antigens from tumor cells, enhancing T-cell infiltration, and directly killing tumor cells. Therefore, this study aims to investigate the efficacy and safety of stereotactic radiotherapy combined with PD-1 inhibitors and chemotherapy in the neoadjuvant treatment of TNBC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed TNBC (ER-, PR-, HER2-)
* 2. cT1cN1-2M0 or cT2N0-2M0；（AJCC 7th）
* 3. ECOG performance status of 0-1;
* 4. Adequate bone marrow function, defined as: Hb ≥ 9.0 g/dL (90 g/L); ANC ≥ 1,500/mcL (1.5 × 10^9/L); PLT ≥ 100,000/mcL (100 × 10^9/L) and no blood transfusion within 3 weeks or growth factor (G-CSF, EPO) therapy within 2 weeks prior to dosing;
* 5. Adequate liver function, defined as: TBIL ≤ 1.5× upper limit of normal (ULN); If no liver metastases, AST and ALT ≤ 2.5× ULN; if liver metastases are present, AST or ALT ≤ 3.0× ULN; ALP ≤ 1.5× ULN; if liver metastases ≤ 2× ULN; Serum albumin ≥ 30g/L;
* 6. Adequate coagulation function: INR or PT, APTT ≤ 1.5× ULN. Participants on anticoagulant therapy should have these laboratory indices closely monitored;
* 7. Adequate renal function, defined as creatinine ≤ 1.5× ULN or Ccr ≥ 50 mL/min calculated using the Cockcroft-Gault formula corrected for body surface area;
* 8. Baseline left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram (ECHO);
* 9. No severe organic heart disease or arrhythmias;
* 10. Women of childbearing potential (aged 15-49 years) must have a negative pregnancy test within 7 days before starting treatment. Both male and female participants of reproductive potential must agree to use effective contraceptive measures during the study period and for 3 months after discontinuation of treatment;
* 11. Voluntary signed informed consent by the study participant.

Exclusion Criteria:

* 1. Patients with a history of mental illness or those diagnosed with mental disorders at the time of enrollment in the clinical trial.
* 2. Patients with communication barriers due to confusion, aphasia, intellectual disability, or other reasons that prevent them from responding normally.
* 3. Poorly controlled tumor-related pain.
* 4. Patients participating in other clinical studies simultaneously.
* 5. Patients with active or past autoimmune diseases or immunodeficiencies, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis.
* 6. A history of idiopathic pulmonary fibrosis, organizing pneumonia (such as obliterative bronchiolitis), drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on chest CT scans at screening.
* 7. Active pulmonary tuberculosis.
* 8. Severe cardiovascular diseases occurring within 3 months prior to the start of study treatment (e.g., NYHA class II or higher heart disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmias, or unstable angina.
* 9. Patients who underwent significant surgical procedures, other than diagnostic surgeries, within 4 weeks prior to the start of the study treatment, or are expected to require significant surgical procedures during the study period.
* 10. Patients who had malignant tumors other than breast cancer within the last 5 years, except for malignancies in the study that have negligible risks of metastasis or death (e.g., a 5-year overall survival rate > 90%), such as adequately treated cervical carcinoma in situ, non-melanoma skin cancer, ductal carcinoma in situ, or stage I uterine cancer.
* 11. Patients who experienced severe infections within 4 weeks prior to the start of the study treatment, including but not limited to those requiring hospitalization due to infections, bacteremia, severe pneumonia, or any active infection that may impact patient safety.
* 12. Patients who have previously received allogeneic stem cell or solid organ transplants.
* 13. Any other diseases, metabolic dysfunctions, physical examination abnormalities, or clinical laboratory abnormalities that contraindicate the use of the study drug, may affect the interpretation of results, or pose a high risk of treatment complications for the patient.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
pCR | The time immediately after the complete surgery
  The percentage of patients showing no evidence of invasive cancer cells in the tissue samples after treatment

SECONDARY OUTCOMES:
Breast conservation rate | 3 year
  The percentage of patients undergoing breast-conserving surgery
Ipsilateral breast recurrence or local regional recurrence | 3 year
  The percentage of patients experiencing a recurrence of cancer in the same breast or in the nearby lymph nodes
Overall survival | 3 year
  The period from the start of treatment until the occurrence of death.
The incidence of adverse events | Up to approximately 1 year
  The safety

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Sichuan, Chengdu, China